CLINICAL TRIAL: NCT04605549
Title: A Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, and Effectiveness of CIN-107 for the Management of Blood Pressure in Patients With Primary Aldosteronism
Brief Title: A Study of CIN-107 in Adults With Primary Aldosteronism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-122; D6970C00001 (Other: AstraZeneca)
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Primary Aldosteronism; Hyperaldosteronism
Keywords: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CIN-107 for dosing at 2, 4, or 8 mg (QD) (Experimental): Patients will be provided with an initial dose of CIN-107 and start once daily (QD) dosing of CIN-107 tablets at 2 mg. At Visit 4, CIN-107 dose may be up-titrated to 4 mg QD if the patient has tolerated dosing of CIN-107 at 2 mg and the blood pressure (BP) records indicate minimal hypotension risk.
  At Visit 5, CIN-107 dose may be up-titrated to 8 mg QD if the patient has tolerated dosing of CIN-107 at 4 mg.
  Interventions: Drug: CIN-107 2 mg dosing; Drug: CIN-107 4 mg dosing; Drug: CIN-107 8 mg dosing

INTERVENTIONS:
Drug: CIN-107 2 mg dosing — One tablet of CIN-107 2 mg tablets, once daily, by mouth, for dosing at 2 mg.
Drug: CIN-107 4 mg dosing — Two tablets of CIN-107 2 mg tablets, once daily, by mouth, for dosing at 4 mg.
Drug: CIN-107 8 mg dosing — Four tablets of CIN-107 2 mg tablets, once daily, by mouth, for dosing at 8 mg.

SUMMARY:
This is a multicenter, open-label study in adult patients with PA to evaluate the effectiveness and safety of CIN-107 after up to 12 weeks of treatment (Part 1), and then for eligible, consenting patients follow patients in Part 2 for up to 74 weeks for evidence of long-term safety and tolerability.

DETAILED DESCRIPTION:
For patients in Part 1 only :

The treatment duration for patients who complete all 3 dose levels, and who opt not to continue in the extension part of the study, is 12 weeks. For patients who do not complete up-titration, the treatment duration will include at least 4 weeks of dosing with the final dose level. If down-titration of CIN-107 dose is determined at Visit 6 (Week 9), the total treatment duration may be extended to 13 weeks to allow sufficient time for CIN-107 treatment effect at the final dose to be assessed. If the final dose of CIN-107 is reached before week 8 (Visit 5) and no up-titration occurs at Visit 5, the patients will be encouraged to continue CIN-107 treatment till Visit 7 for a total of 12 weeks of treatment. The patients who opt not to continue to Part 2 will not receive any study drug and will return for their safety follow up visit (Visit 8) in 2 weeks.

For patients who opt to continue in the extension part (Part 2) of the study:

Patients will continue to receive their dose of baxdrostat and be instructed to measure BP at least once every week prior to dosing with CIN-107 in the morning, during the extension phase. Safety surveillance will be conducted if clinically indicated. Repeat and unscheduled testing for serum potassium may be measured at the investigator's clinical site or at local laboratory for a faster turn-around time to allow clinical assessment. These patients entering part 2 will skip Visit 8 and their next visit will be Visit 9.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with PA.
2. Are taking mineralocorticoid receptor antagonist (MRA) to control BP; or are newly diagnosed with PA and have not started MRA treatment.
3. Are willing and able to cease dosing of MRA for up to 4 weeks in patients taking MRA.
4. Are willing to be compliant with the contraception and reproduction restrictions of the study.
5. Have increased SBP by ≥ 20 mmHg or have SBP ≥ 160 mmHg after dosing of MRA treatment is ceased for up to 4 weeks duration, or have SBP ≥ 150 mmHg for patients who are newly diagnosed with PA and have not taken an MRA in the past 12 weeks.

Exclusion Criteria:

1. At Screening Visit, have a single occurrence of mean seated SBP > 180 mmHg or DBP > 110 mmHg if not taking an MRA; or have a mean seated SBP ≥ 160 mmHg or DBP ≥ 100 mmHg if currently taking an MRA.
2. Have a body mass index > 45 kg/m2.
3. Have had a previous surgical intervention for an adrenal adenoma or have a planned adrenal carcinoma, adrenalectomy, renal nerve denervation, or adrenal ablative procedure during the course of the study.
4. Have a documented estimated glomerular filtration rate < 45 mL/min/1.73 m2.
5. Have a planned dialysis, kidney transplantation or any major surgical procedure during the course of the study.
6. Have known documented New York Heart Association class III or IV chronic heart failure.
7. Have had a stroke, transient ischemic attack, hypertensive encephalopathy, acute coronary syndrome, or hospitalization for heart failure within 6 months before the Screening Visit.
8. Have known current severe left ventricular outflow obstruction.
9. Have had major cardiac surgery within 6 months before the Screening Visit.
10. Have a history of, or currently experiencing, clinically significant arrhythmias.
11. Have had a prior solid organ transplant or cell transplant.
12. Are positive for HIV antibody, hepatitis C virus RNA, or hepatitis B surface antigen.
13. Have typical consumption of > 14 alcoholic drinks weekly.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CIN-107 | 74 Weeks
  Outcome measure is overall safety with is a composite of the following individual parameters (unit of measure in brackets):
  * Adverse Events [number of events];
  * ECGs [PR interval (msec), RR interval (msec), or QTcF interval (msec); clinically significant ECG findings that are detected during the study will be reported as adverse events];
  * Clinical laboratory evaluations including standard safety chemistry panel, hematology, coagulation, and urinalysis [clinically significant abnormal laboratory findings that are detected during the study will be reported as adverse events];
  * Vital signs [pulse, temperature, heart rate and blood pressure] and physical examination data changes noted as clinically significant abnormalities that arise during the study will be recorded as adverse events
Change in mean seated systolic blood pressure (SBP) | after 12 weeks of treatment
  Effectiveness measured by change in mean seated SBP after 12 weeks of treatment in patients with PA

SECONDARY OUTCOMES:
Change in mean diastolic blood pressure (DBP) | after 12 weeks of treatment
  Comparison of changes in mean SBP after 12 weeks of treatment in patients with PA.
The percentage of patients achieving a seated blood pressure (BP) response <140/90 mmHg | at Week 12
  The percent of patients who achieved a seated BP response <140/90 mmHg after CIN107 treatment will be evaluated at each dose level at Week 12.
The percentage of patients achieving a seated BP response <130/80 mmHg | at Week 12
  The percent of patients who achieved a seated BP response <130/80 mmHg after CIN107 treatment will be evaluated at each dose level at Week 12.
The percentage of patients achieving either: - a plasma aldosterone concentration (PAC) < 15 ng/dL and a plasma renin activity (PRA) ≥ 0.5 ng/mL/h; or - an ARR < 15; or - unsuppressed renin activity PRA ≥ 1.0 ng/mL/h | after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Greenbrae, California
  - Research Site, San Francisco, California
  - Research Site, West Hollywood, California
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Townsend RR. Blocking Aldosterone Synthesis: Whose BrigHTN Idea Was That? Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1631-1633. doi: 10.2215/CJN.0000000000000265. Epub 2023 Jul 24. No abstract available. PMID 37490693